CLINICAL TRIAL: NCT07199608
Title: A Combined Subcision Approach With Either Fractional CO₂ Laser or Platelet-rich Plasma Versus Subcision Alone in the Treatment of Atrophic Post-acne Scars
Brief Title: Subcision With CO₂ Laser or PRP vs Subcision Alone in Atrophic Acne Scars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmeen Gamal Abdel Halim Ahmed, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: subcision in acne scars
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Atrophic Acne Scar

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- subcision alone (Active Comparator)
  Interventions: Procedure: subcision
- subcision+fractional co2 laser (Experimental)
  Interventions: Procedure: subcision+fractional co2 laser
- subcision+platelet rich plasma (Experimental)
  Interventions: Biological: subcision+PRP

INTERVENTIONS:
Procedure: subcision — patients will undergo subcision procedure alone using 18 gauge blunt cannula to release fibrous bands under atrophic acne scars.this group will serve as control comparator
  Arms: subcision alone
Procedure: subcision+fractional co2 laser — patients will undergo subcision procedure followed by fractional co2 laser applied to right side of face, the left side will receive subcision alone
  Arms: subcision+fractional co2 laser
Biological: subcision+PRP — patients will undergo subcision procedure followed by intradermal injection of autologous PRP prepared from patients blood on right side.left side will receive subcision alone
  Arms: subcision+platelet rich plasma

SUMMARY:
Acne vulgaris is an inflammatory disease of pilosebaceous unit ,leading to different types of scars including atrophic, hypertrophic and keloidal. Atrophic scars are the most common type ,affecting about 75-90% of acne scar cases and can be ice pick, rolling or boxcar in morphology . Theses scars may cause significant impact such as depression, anxiety , and reduced quality of life. multiple treatment modalities exist, including lasers ,chemical peels, dermabrasion, microneedling, subcision and platelet rich plasma. Subcision is a well established technique that improves rolling and boxcar scars by releasing fibrotic strands. Fractional co2 laser induces dermal remodeling and collagen neogenesis, while PRP enhances wound healing and collagen induction through growth factors. Combinig subcision with either co2 laser or PRP may enhance treatment efficacy compared to subcision alone.

rational : Subcision alone may provide limited improvement in some patients. Fractional CO₂ laser and PRP are promising adjunctive modalities that could enhance collagen remodeling and improve cosmetic outcomes. Evaluating their combined effect versus subcision alone will help determine the most effective and safe approach for managing atrophic post-acne scars.

aim of work:To compare the efficacy and safety of combined subcision with either fractional CO₂ laser or platelet-rich plasma versus subcision alone in the treatment of facial atrophic post-acne scars.

DETAILED DESCRIPTION:
Type of the study: Prospective, comparative, split-face study. - Study Setting: The study will be done in Assiut University Hospital ,dermatology department ,after obtaining approval from ethics committee of Faculty of Medicine, Assiut University in Assiut, Egypt.

Sample Size Calculation:

Based on determining the main outcome variable, the estimated minimum required sample size is 42 cases (21 in each group). Sample size was calculated using G*Power software version 3.1.9.7, based on the following assumptions: The main outcome is the difference in mean Goodman and Baron quantitative scar score between two independent groups of patients: those treated with Subcision + PRP and those treated with Subcision + Fractional CO₂.

Based on clinical experience and after reviewing the literature, a large difference was assumed.

The main statistical test is a one-tailed independent t-test to detect the difference between two means.

Effect size = 0.8 Alpha = 0.05 Power = 0.80

All patients will undergo subcision on both sides of the face, patients will be randomly divided into two groups:

group I (21 patients)-subcision combined with platelet rich plasma injection at right side of the face and subcision alone at the other side.

group II (21 patients)-subcision combined with fractional CO2 at right side of the face and subcision alone at the other side .

Each side will be randomly selected by choosing a sealed opaque envelope containing a card labeled with either laser or PRP representing the right split face side treatments.

Each patient will undergo three sessions with one month interval in between. Patient preparation

1. Each patient's entire face will be disinfected with alcohol and cleaned with saline.
2. Anesthesia will be injected subcutaneously with 2% lidocaine
3. A sharp needle inserted at a shallow angle, with the blade facing upward, at the periphery of the scarred area to create a pathway to facilitate the entry of the blunt cannula.
4. Subcision will be performed with an 18-gauge blunt cannula introduced at a 30° angle into the mid to deep dermis, then moved back and forth in a fan-like motion under the scar to release fibrous bands at the dermal or deep dermal, subcutaneous plane until the sound of bands breaking lost, and no resistance felt (endpoint).
5. To establish hemostasis, firm pressure should be applied for at least 5 min.
6. After subcision, the face should be cleaned with alcohol swabs and then sterile saline.

PRP side (group I): Right side of the face will be injected with PRP and the other by saline.

Fractional side (group II): Right side of the face will be treated with a fractional CO2 laser (10,600 nm) using post acne scar mode (DAESHIN ENTERPRISE CO2, LTD. (D.S.E) 105,207,Digital ro,Guro-gu, Seol, Korea).

Post procedure care All patients should be instructed to avoid sunlight exposure and to use sunscreen (SPF ≥ 50).

Cold compresses in first 24h-48h to avoid edema and ecchymosis. Use topical antibiotic ointment as mupirocin or fusidic acid. Analgesics as paracetamol to decrease the pain.

-Research outcome measures:

1. Primary (main):

   Goodman & Baron qualitative & quantitative grading systems.
2. Secondary (subsidiary):

Photography, quartile grading scale. dermoscopic evaluation (erythema, pigmentation, photodamage, follicular density) Data entry and analysis will be carried out using SPSS version 21. Descriptive statistics will be performed with frequency and percentages for categorical variables. Mean and standard deviation for normally distributed numerical variables, while median and interquartile measures for non-normally distributed numerical. Then analytic statistics will be done as the chi-square test for comparing independent categorical variables, and McNemar's test. If the data is normally distributed independent t-test, paired t-test, ANOVA, and Pearsons correlations tests will be used. If the data is not normally distributed Mann-Whitney, Kruskal-Wallis, Willcoxon signed-rank, Friedman, and Spearmans correlation tests will be used. Values will be considered significant when P values equal or less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* - Adult patients of both sexes with mild to severe atrophic post-acne scars.

Exclusion Criteria:

* - Age < 18 years
* Pregnant or lactating women
* Active inflammatory acne or infection in treatment area
* Premalignant or malignant lesions
* Photosensitive dermatoses
* Coagulation defects or blood disease
* History of keloid scars
* Systemic retinoid use in previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Goodman and Baron quantitative acne scar score (Baseline vs 1 month post last session). | 3 sessions per patient at 1-month intervals Follow-up: 1 month after last session
  If the scale was lowered by: (Quantitative) 0-5 points, the reduction will be considered minimal 5-10 points, it will be considered moderate reduction 10-15 points, it will be considered good reduction >15 points, it will be considered very good reduction

SECONDARY OUTCOMES:
Quartile grading scale improvement - Dermoscopic evaluation (erythema, pigmentation, photodamage, follicle density) | 3 sessions per patient at 1-month intervals Follow-up: 1 month after last session
  0 = slight improvement if <25%
  1. = moderate improvement if 25-49%
  2. = significant improvement if 50-74%
  3. = marked improvement if >75

CONTACTS AND LOCATIONS:
Overall Officials: Azza Mahfouz Abdel Meguid, Study Chair — Assiut University; Reham Maher Abd El Gaber, Study Director — Assiut University
Locations (1):
- Assiut University Hospitals, Dermatology Department, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Tran BQ, Tran TNA, Doan EVL, Nguyen TTP, Nguyen HT. Simultaneous versus sequential fractional CO2 laser and subcision combination for management of post-acne atrophic scars: A split-face comparative study. J Cosmet Dermatol. 2024 Oct;23(10):3210-3221. doi: 10.1111/jocd.16395. Epub 2024 May 21. PMID 38770894
- [Background] Abdelwahab AA, Omar GAB, Hamdino M. A combined subcision approach with either fractional CO2 laser (10,600 nm) or cross-linked hyaluronic acid versus subcision alone in atrophic post-acne scar treatment. Lasers Med Sci. 2022 Dec 24;38(1):20. doi: 10.1007/s10103-022-03677-y. PMID 36564573
- See also: Related Info — https://link.springer.com/